CLINICAL TRIAL: NCT03942705
Title: A New Approach to Cervical Cancer Prevention in Kenya
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Academic Model Providing Access to Healthcare (AMPATH) (Other)
Responsible Party: Principal Investigator, Darron Brown MD, MPH, Professor of Medicine, Indiana University
Other Study IDs: 1712513308
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: human papillomavirus (HPV); cervical cancer; prevention; Kenya
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervico-vaginal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kenyan Women: Women living in western Kenya will be asked to complete a self collected vaginal sample for HPV DNA screening and asked to undergo a second screening by VIA. As per Kenyan standard of care, vaccination against HPV will be offered to children/grandchildren (boys and girls) of women, and to the women themselves if age 26 or younger. The second vaccine dose (for children ages 9 through 14) and third doses (for children and adult women ages 15 through 26) will be administered at subsequent visits. There will be no requirement for HPV vaccination (of children or mothers up to 26 years of age) for participation in the study. Results of the screening will be returned to participants and they will be referred to receive standard care as applicable.

SUMMARY:
The purpose of this study is to determine if the human papillomavirus (HPV) deoxyribonucleic acid (DNA) testing, performed on self-collected vaginal swabs, is acceptable, feasible, and sensitive and specific in detection of high-grade cervical lesions among Kenyan women, compared to the current standard of care.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that effective cervical cancer screening can be performed in a high percentage of women, using HPV DNA of self-collected vaginal samples, provided by women attending either chamas (community groups) or in their own homes. HPV DNA testing will be used to triage women for a secondary screen by visual inspection with acetic acid (VIA) in a local clinic. The investigators will determine if HPV DNA testing, performed on self-collected vaginal swabs, is acceptable, feasible, and sensitive and specific in detection of high-grade cervical lesions among Kenyan women, compared to the current standard of care. In addition, women will bring their children to be vaccinated against HPV in these community meetings, using the standard of care for the approved HPV vaccine available in Kenya.

The investigators will test this approach by completing the following Specific Aims:

Specific Aim 1: Determine the percentage of women attending community meetings who will provide self-collected vaginal swabs for HPV DNA testing.

Specific Aim 2. Following HPV DNA screening using self-collected swabs, determine the percentage of these women who will attend the local clinic.

Specific Aim 3. Evaluate the statistical correlation between HPV DNA testing of self-collected vaginal swabs and VIA (as all women in this pilot study will undergo VIA).

ELIGIBILITY:
Inclusion Criteria:

1. Women who live in Kenya who are between the ages of 30 and 55, are willing to provide a self collected vaginal swab and willing to travel to the local clinic for a VIA

Exclusion Criteria:

1. current pregnancy, inability to consent due to mental or physical disability, or a medical illness that has rendered the patient unable to understand consent

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Kenyan women between the ages of 18 and 60 who are willing to provide a self-collected vaginal swabs and willing to travel to the local clinic for VIA.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of women attending community meetings who will provide self-collected vaginal swabs for HPV DNA testing. | anytime after informed consent up to 2 years
Percentage of women who attend clinic after providing self-collected vaginal swabs | any time after completion of self-collected vaginal swab (up to 2 years)

SECONDARY OUTCOMES:
HPV DNA vaginal swab testing results | any time after after self-collected vaginal swab, up to 2 years
  analyzed for the human reference gene (specimen adequacy), HPV 16/18, or any of 12 oncogenic HPV types.
Visual inspection with acetic acid (VIA) testing results | any time after VIA is performed, up to 2 years
  Results reported as abnormal or normal

CONTACTS AND LOCATIONS:
Overall Officials: Darron Brown, MD, Principal Investigator — Indiana University
Locations (1):
- Moi University, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available after deidentification. Other documents including study protocol, statistical analysis plan, informed consent form, case study reports, will also be available. These documents will be available beginning three months after publication, and will end 12 months following publication. Data will be available to researchers who provide a methodologically sound proposal. Proposals should be directed to darbrow@iu.edu. To gain access, data requesters will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 to 12 months
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal.